CLINICAL TRIAL: NCT00058851
Title: Massage Therapy for Breast Cancer-Related Lymphedema
Brief Title: Massage Therapy for Breast Cancer Treatment-Related Swelling of the Arms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT001326-01 (NIH)
Record Dates: First submitted 2003-04-14; First posted 2003-04-15 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Lymphedema
Keywords: Manual lymph drainage; Combined physiotherapy
MeSH Terms: conditions — Lymphedema | interventions — Manual Lymphatic Drainage; Compression Bandages

INTERVENTIONS:
Procedure: Manual lymph drainage
Procedure: Combined physiotherapy
Procedure: Compression bandaging

SUMMARY:
The purpose of this study is to examine the short-term and long-term efficacy of massage therapy alone compared to massage therapy plus compression bandaging in the treatment of breast cancer treatment-related swelling of the arms and legs.

DETAILED DESCRIPTION:
Massage therapy (in the form of manual lymph drainage [MLD]) and compression bandaging (CB) are integral components of combined physical therapy (CPT), the recommended treatment for peripheral lymphedema (LE). According to the World Health Organization, LE afflicts hundreds of millions worldwide and probably millions in the United States. Effects of various forms of massage on lymph circulation have been postulated for more than a century, but the efficacy of MLD alone without CB has not been demonstrated. New data suggest that MLD alone reduces established LE volume as effectively as CB in combination with CPT and minimizes LE development.

Patients will be randomly assigned to either treatment with MLD alone or a combination of MLD and CB. Patients will be treated in 10 one-hour sessions over 2 weeks. They will also undergo lymphangioscintigraphy (a nuclear medicine test) to depict the function of their lymphatic system. Patients will continue self treatment at home and will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Lymphedema (5% to 20% increase in volume) after breast cancer treatment

Exclusion Criteria:

* Physically unable to perform massage or bandaging during home program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2003-01; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
volume change

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bernas, MS, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States